CLINICAL TRIAL: NCT01922141
Title: A Randomized, Double-blind, Parallel Group, Active-controlled Study to Compare the Systolic Blood Pressure Lowering Efficacy of Aliskiren, Ramipril and a Combination of Aliskiren and Amlodipine, With an Initial 8-week Evaluation, Followed by a 2-3 Year Follow-up to Compare Long-term Safety of an Aliskiren-based Regimen to a Ramipril-based Regimen in Hypertensive Patients ≥ 65 Years of Age
Brief Title: Aliskiren Study of Safety and Efficacy in Senior Hypertensives
Acronym: ASSESS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPP100A2370; 2013-001562-42 (EudraCT Number)
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension
Keywords: High blood pressure, stage 1 and 2 hypertension
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Amlodipine; Ramipril; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aliskiren monotherapy (Experimental): Aliskiren 150 mg, once a day, force titrated to Aliskiren 300 mg after 8 weeks in 50% of patients. Optional addition/titration of amlodipine 5 mg/10 mg and hydrochlorothiazide 12.5/25 mg based on systolic BP control in sequential steps
  Interventions: Drug: Aliskiren; Drug: Amlodipine; Drug: Hydrochlorothiazide
- Aliskiren dual therapy (Experimental): Aliskiren 150 mg plus amlodipine 5 mg, once a day, force titrated to Aliskiren 300 mg plus amlodipine 5 mg after 8 weeks in 50% of patients. Optional titration of amlodipine 5 mg to 10 mg and optional addition/titration of hydrochlorothiazide 12.5/25 mg based on systolic BP control in sequential steps
  Interventions: Drug: Aliskiren; Drug: Amlodipine; Drug: Hydrochlorothiazide
- Ramipril monotherapy (Active Comparator): Ramipril 5 mg, once a day, force titrated to Ramipril 10 mg after 8 weeks in 50% of patients. Optional addition/titration of amlodipine 5 mg/10 mg and hydrochlorothiazide 12.5/25 mg based on systolic BP control in sequential steps
  Interventions: Drug: Amlodipine; Drug: Ramipril; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 mg and aliskiren 300 mg tablets will be supplied centrally. These will be blinded with matching placebos for the 2 dose strengths.
  Other Names: Rasilez, Tekturna
  Arms: Aliskiren dual therapy; Aliskiren monotherapy
Drug: Amlodipine — Amlodipine 5 mg/10 mg will also be blinded and supplied centrally. For Aliskiren dual therapy arm , Amlodipine is in the regimen; where as for monotherapy arms, Amlodipine is an optional add-on therapy.
Drug: Ramipril — Ramipril 5 mg and ramipril 10 mg capsules will be supplied centrally. These will be blinded with matching placebos for the 2 dose strengths.
  Arms: Ramipril monotherapy
Drug: Hydrochlorothiazide — Hydrochlorothiazide 12.5 mg/25 mg will be open label and supplied locally. It is an optional add-on to each arm.

SUMMARY:
This study is designed to compare the blood pressure lowering efficacy of aliskiren, a combination of aliskiren plus amlodipine, and ramipril in elderly patients with mild to moderate hypertension. It will also compare the long-term safety of an aliskiren-based regimen to a ramipril-based regimen

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 65 years of age with a clinical diagnosis of essential hypertension at Visit 1.
* Mean sitting SBP (MSSBP) ≥ 140 mmHg and < 180 mmHg at Visit 2/Visit 201 and Visit 3.
* Absolute MSSBP difference ≤ 20 mmHg between Visit 3 and the Visit immediately prior

Exclusion Criteria:

* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
* Severe hypertension (MSSBP ≥ 180 mmHg or MSDBP ≥ 110 mmHg) at Visit 1, Visit 2, Visit 201 or Visit 3 or during patient self measured blood pressure (SMBP) monitoring in the pre-randomization period confirmed by office measurement.
* Current treatment with any blocker of the renin angiotensin aldosterone system (RAAS) (aliskiren, ACE inhibitor, angiotensin receptor blocker or an aldosterone antagonist) and unable to discontinue this therapy.
* Concurrent use of any anti-hypertensive medications except a stable dose of 3 months prior to Visit 1 of alpha adrenergic blockers for benign prostatic hypertrophy (e.g., tamsulosin [Flomax®] for benign prostatic hypertrophy), beta blockers for angina, or beta blocker ophthalmic preparations.
* Contraindications to aliskiren, ramipril, amlodipine, or hydrochlorothiazide. Other protocol defined inclusion/exclusion criteria apply

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure (MSSBP) to week 8 | Baseline, Week 8
  The change from baseline to week 8 in mean sitting systolic blood pressure will be analyzed for aliskiren monotherapy, dual therapy of aliskiren and amlodipine and ramipril monotherapy using ANCOVA model in which treatment arm, region and age (less than 75 and greater than or equal to 75 years) will be included as factors

SECONDARY OUTCOMES:
Number of patients with serious adverse events and adverse events | Baseline, Week 8, average 2.5 years
  Safety and tolerability of study treatments will be analyzed by comparing the frequency of serious adverse events and adverse events at the time frames
Number of patients with hyperkalemia, hypotension and reduction of estimated glomerular filtration rate (eGFR) | Baseline, Week 8
  The incidence of hyperkalemia, hypotension and reduction of eGFR will be compared between aliskiren monotherapy, aliskiren dual therapy with amlodipine and ramipril monotherapy
Change from baseline in mean sitting systolic blood pressure (MSSBP) at the end of double blind period | Baseline, end of double blind period (in average 2.5 years)
  Change in mean sitting systolic blood pressure will be analyzed for the aliskiren-based regimen vs. the ramipril based regimen
Percentage of patients achieving blood pressure control | Baseline, Week 8, average 2.5 years
  Percentage of patients achieving blood pressure control, defined as mean sitting systolic BP below 140 mmHg and mean sitting diastolic BP below 90 mmHg, will be analyzed for the study treatments
Percentage of patients with major cardiovascular events | Average 2.5 years
  Percentage of patients with major cardiovascular events (defined as composite of cardiovascular death, resuscitated cardiac death, non-fatal stroke, non-fatal myocardial infarction, heart failure hospitalization and atrial fibrillation) will be analyzed for the aliskiren-based regimen and the ramipril-based regimen
Number of patients with gastrointestinal tract cancer | Average 2.5 years
  The frequency of gastrointestinal tract cancer (malignant neoplasms of mouth, esophagus, stomach, small intestine, appendix, anus, gastrointestinal stroma, colon and rectum, excluding pancreatic, biliary tract and liver cancers) will be analyzed for the aliskiren-based regimen and the ramipril-based regimen

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals